CLINICAL TRIAL: NCT02156362
Title: Determination of Pronostics Factors for Advanced Thyroid Carcinoma (pT3 pT4 or M1 at Diagnosis)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011.665
Record Dates: First submitted 2012-05-29; First posted 2014-06-05 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Thyroid Cancer
Keywords: Thyroid carcinoma; predictive factors; refractory; Differentiated; follicular origin
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- follow up (Other)
  Interventions: Other: follow up visit

INTERVENTIONS:
Other: follow up visit — At least 1 follow up visit per year will be done and an additional visit if needed.

SUMMARY:
It is generally estimated that 5 % of patients with thyroid cancer will develop distant metastases, and most of them had an advanced stage of the disease at presentation. Thirty per cent of them are resistant to radio iodine therapy and are called "refractory". Their long term survival is estimated to be less than 10 %.

The objective of this study is to identify the factors associated with poor outcome in a cohort of patients with advanced thyroid cancer followed during 5 years. Anaplastic and medullary thyroid carcinomas were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥ 18 years.
* Thyroid cancer differentiated from follicular origins (papillary, vesicular or poorly differentiated carcinoma).
* TNM classification: stage pT3 (≥2 cm), or pT4 or M1 at diagnosis.
* Patient after post operative radioiodine therapy.

Exclusion Criteria:

* Patient who can not be followed during the protocol.
* Patient who does not consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Estimated)
Dates: Start 2012-05 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Rate of Thyroid cancer evolving to refractory stage | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Claire BOURNAUD, MD, Principal Investigator — Hospices Civils de Lyon- Centre de Médecine Nucléaire Groupement hospitalier est, 59 boulevard Pinel, 69677 Bron cedex
Locations (1):
- Hospices Civils de Lyon-Centre de Médecine Nucléaire Groupement Hospitalier Est 59 boulevard Pinel, Bron, France